CLINICAL TRIAL: NCT04257461
Title: BALLAD BELGIUM: A Trial to Evaluate the Potential Benefit of Adjuvant Chemotherapy for Small Bowel Adenocarcinoma
Brief Title: A Trial to Evaluate the Potential Benefit of Adjuvant Chemotherapy for Small Bowel Adenocarcinoma
Acronym: BALLAD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Belgian Group of Digestive Oncology (Other)
Collaborators: Kom Op Tegen Kanker (Other); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BALLAD BELGIUM
Record Dates: First submitted 2020-01-09; First posted 2020-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-02

CONDITIONS: Small Bowel Adenocarcinoma
MeSH Terms: interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group1 Arm A (No Intervention): Observation only
- Group 1 Arm B (Other): Mono- or bichemotherapy: fluoropyrimidine with or without Oxaliplatin (choice by physician/patient or by randomisation)
  Interventions: Drug: Fluoropyrimidine; Drug: Oxaliplatin
- Group 2 Arm C (Other): Monochemotherapy: fluoropyrimidine
  Interventions: Drug: Fluoropyrimidine
- Group 2 ARM D (Other): Bichemotherapy: fluoropyrimidine with oxaliplatin
  Interventions: Drug: Fluoropyrimidine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Fluoropyrimidine — Monotherapy: 12 cycles of 5FU or 8 cycles of Capecitabine. The choice of fluoropyrimidine must be specified prior to randomisation.
  Other Names: Capecitabine; LV5FU2
  Arms: Group 1 Arm B; Group 2 ARM D; Group 2 Arm C
Drug: Oxaliplatin — Bichemotherapy: Oxaliplatine combined with Fluoropyrimidine.
  Other Names: Xeloda
  Arms: Group 1 Arm B; Group 2 ARM D

SUMMARY:
An open-label, randomised, controlled, multi-centre, trial with disease free survival as the primary end point. The worldwide collaboration is referred to as GLOBAL BALLAD and consists of a number of individual parallel prospective studies addressing the same objectives with similar designs brought together under the framework of the International Rare Cancer Initiative. This protocol is for BALLAD BELGIUM, which is the component of GLOBAL BALLAD.

DETAILED DESCRIPTION:
The utility of adjuvant chemotherapy in the management of Small Bowel Adenocarcinoma (SBA) remains unproven and awaits the results of a large, global, prospective, phase III, randomised, controlled trial. Across the 830 million population of North America and Europe, there are approximately 3,000 patients with R0 resected and potentially cured SBA every year who would be potentially eligible for such an adjuvant chemotherapy trial.

Given the absence of good-quality and evidence-based data, it has been agreed that a trial considering adjuvant chemotherapy versus no chemotherapy was appropriate for patients with stage I-IV SBA in whom the oncologist and patient feel that the benefit of adjuvant chemotherapy is uncertain. For those patients with stage I-IV SBA who, with their oncologists, feel that the potential benefit of adjuvant chemotherapy is certain (and hence are not willing to accept randomisation to the 'no chemotherapy' arm), a randomisation between single agent fluoropyrimidine versus doublet fluoropyrimidine and oxaliplatin chemotherapy will be offered. Tumour stage will be used as a stratification factor. Those patients who do not consent to be randomised will be offered registration to allow collection of demographic, clinicopathological, epidemiological and survival data, thereby making optimal use of the rare patient population available. In addition, archival Formalin Fixed Paraffin Embedded (FFPE) tissue and contemporaneous venous blood samples will be collected from every registered patient to allow molecular profiling and future translational research. A questionnaire about underlying risk factors (e.g. Crohn's disease, coeliac disease, Lynch syndrome etc) will be completed along with the other collected data on all registered patients.

The trial hypotheses are that:

1. Adjuvant chemotherapy results in an improved outcome (DFS and OS) over observation alone after potentially curative R0 surgery for stage I, II, III and IV SBA
2. Adjuvant fluoropyrimidine and oxaliplatin chemotherapy results in an improved outcome (DFS and OS) over fluropyrimidine alone after potentially curative R0 surgery for stage I, II, III and IV SBA.

ELIGIBILITY:
Inclusion Criteria:

1. R0 resected stage I, II or III SBA
2. No evidence of residual or metastatic disease at laparotomy and on CT/MRI imaging of chest, abdomen and pelvis.
3. Patients must be registered and randomised within 12 weeks of surgery and commence chemotherapy within 14 weeks of surgery
4. ECOG Performance Status of 0 or 1
5. Absolute neutrophil account ≥ 1.5 x109/l
6. Platelet count ≥ 100 x 109/l
7. Haemoglobin ≥90 g/l (previous transfusion is allowed)
8. AST and ALT ≤ 2.5 x upper limit of normal (ULN). (At least one of ALT or AST MUST be performed)
9. Creatinine clearance > 50 ml/min (calculated by Cockcroft Gault or Wright equation) or measured by EDTA
10. Serum bilirubin ≤ 1.5 x ULN
11. Signed and dated informed consent indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrolment.
12. Age ≥ 18 years
13. Willingness and ability to comply with scheduled visits, treatment plans and laboratory tests and other trial procedures.

Exclusion Criteria:

1. Non-adenocarcinoma histology of small bowel tumour which includes but is not confined to lymphoma, GIST, carcinoid or other neuroendocrine tumour, squamous carcinoma, melanoma or sarcoma.
2. Previous neo-adjuvant chemo(radio)therapy for SBA
3. Clinically significant cardiovascular disease (i.e. active or < 12 months since cerebrovascular accident, myocardial infarction, unstable angina, New York Heart Association [NYHA] grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, uncontrolled hypertension)
4. Pregnancy/lactation or of child bearing potential and not using medically approved contraception. (Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential)
5. Previous malignancy other than adequately treated in situ carcinoma of the uterine cervix or basal or squamous cell carcinoma of the skin, unless there has been a disease free interval of at least 3 years and treatment was with curative intent
6. Known or suspected dihydropyrimidine dehydrogenase (DPD) deficiency
7. Known untreated coeliac disease (may be enrolled if diet controlled), untreated chronic inflammatory bowel disease or other cause of malabsorption or intestinal obstruction
8. Grade ≥ 2 peripheral neuropathy
9. Administration of any investigational drug within 28 days or 5 halflives, whichever is longer, prior to receiving the first dose of trial treatment.
10. Previous hypersensitivity to platinum salts
11. Patients with clinically significant, active infections, or any other serious medical condition in which chemotherapy is contraindicated will be excluded
12. Patients with untreated vitamin B12 deficiency are excluded from receiving folinic acid as part of their chemotherapy regimen. However, these patients may be eligible for treatment with capecitabine fluoropyrimidine therapy, where no folinic acid is administered as part of the treatment regimen
13. Patients with clinically significant sensorineural hearing impairment are excluded from receiving oxaliplatin but will be eligible for the fluoropyrimidine monotherapy provided as a clinician's choice for patients in group 1 randomised to either observation or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
efficacy assessed by the 3-year Disease-free survival | 3 years from randomisation
  This is defined as time from randomisation to the first occurrence of the following events:
  * Disease relapse (confirmed by imaging)
  * Incidence of a new primary (confirmed by imaging and histology/cytology)
  * Death from any cause

SECONDARY OUTCOMES:
efficacy assessed by the overall survival | 5 years from randomisation
  The patient's survival status is determined at each follow-up visit. After the mandated clinic visits survival status data will come from responsible cancer centres, cancer registries and national databases and include long-term passive follow-up data.
safety assessed by the toxicity of chemotherapy | until 1 month after treatment
  Toxicity will be assessed using CTCAE version 4.0. Only toxicities that are at least grade 2 will be recorded on the CRF
quality of life as assessed using the EORTC (European Organisation for Research and Treatment of Cancer) Quality of Life Questionnaire Core 30 | until end of study, up to 5 years from randomisation
  This will be completed at 9, 12, 18 and 24 months post randomisation for all arms of the trial. Minimum and maximum values do not apply for this scale.
quality of life as assessed using the EORTC (European Organisation for Research and Treatment of Cancer) Quality of Life Questionnaire Colo-Rectal module 29 | until end of study, up to 5 years from randomisation
  This will be completed at 9, 12, 18 and 24 months post randomisation for all arms of the trial. Minimum and maximum values do not apply for this scale.
quality of life as assessed using the EuroQol 5 dimension scale (EQ-5D) | until end of study, up to 5 years from randomisation
  This will be completed at 9, 12, 18, 24, 30, 36, 48, 60 72 and 84 months post randomisation for all arms of the trial. Minimum and maximum values do not apply for this scale.
Exploratory: clinical applicability of the study results assessed by the translational research on blood and tissue | Will be collected at the end of study, up to 5 years from randomisation
  The aim is to establish a biobank of SBA tissue and blood with complete and comprehensive trial quality follow-up data which may act as the foundation for many future collaborative research projects and for combined projects with other funded tissue collections.

CONTACTS AND LOCATIONS:
Overall Officials: Timon Vandamme, Prof, Principal Investigator — Coordinating Investigator
Locations (9):
- Belgium (9):
  - AZ Turnhout, Turnhout, Antwerpen
  - UZ Antwerpen, Antwerp, Antwerp
  - ULB Erasme, Brussels, Brussels Capital
  - Cliniques Universitaires Saint-Luc UCL, Brussels, Brussels Capital
  - CHC MontLégia, Liège, Liège
  - CHU Liège, Liège, Liège
  - Onze-Lieve-Vrouw Ziekenhuis Aalst, Aalst, Oost-Vlaanderen
  - AZ St-Lucas, Ghent, Oost-Vlaanderen
  - AZ Delta, Roeselare, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: No